CLINICAL TRIAL: NCT01316718
Title: Efficacy and Mode of Action of Mesalazine in the Treatment of Diarrhoea-predominant Irritable Bowel Syndrome (IBS-D).
Brief Title: Mesalazine for the Treatment of Diarrhoea-predominant Irritable Bowel Syndrome (IBS-D)
Acronym: MIBS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10085
Record Dates: First submitted 2010-09-21; First posted 2011-03-16 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Irritable Bowel Syndrome With Diarrhoea
Keywords: IBS; diarrhoea
MeSH Terms: conditions — Diarrhea | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesalazine Granules (Experimental): 2g oral granules, once a day for 1 week, then 2g oral granules, twice a day for 11 weeks
  Interventions: Drug: Mesalazine
- Placebo Granules (Placebo Comparator): 2g oral granules, once a day for 1 week, then 2g oral granules, twice a day for 11 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalazine — 2g oral granules, once a day for 1 week, then 2g oral granules, twice a day for 11 weeks
  Arms: Mesalazine Granules
Drug: Placebo — 2g oral granules, once a day for 1 week, then 2g oral granules, twice a day for 11 weeks
  Arms: Placebo Granules

SUMMARY:
The purpose of the trial is to define the clinical benefit and possible mediators of the benefit of mesalazine in Irritable Bowel Syndrome (IBS) with diarrhoea.

The investigators will therefore evaluate symptoms (primarily bowel frequency) and markers reflecting mast cell activation and small bowel tone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients aged 18-75 years old able to give informed consent.
2. Patients should all have had a colonoscopy or a sigmoidoscopy within the last 12 months to exclude microscopic colitis. (If not, but they have had a negative colonoscopy within 5 years and symptoms are unchanged, then a sigmoidoscopy and mucosal biopsy of the left colon would be sufficient to exclude microscopic colitis).
3. IBS-D Patients meeting Rome III criteria prior to screening phase.
4. Patients with ≥ 25% soft (score > 4) and < 25% hard (score 1 or 2) stools during the screening phase, as scored by the daily symptom and stool diary*.
5. Patients with a stool frequency of 3 or more per day for 2 or more days per week during the screening phase*.
6. Satisfactory completion of the daily stool and symptom diary during the screening phase at the discretion of the investigator.
7. Women of child bearing potential willing or able to use at least one highly effective contraceptive method throughout the study. In the context of this study, an effective method is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly such as: implants, injectables, combined oral contraceptives, sexual abstinence or vasectomised partner.

   * If inclusion criterion 4 and/or 5 is/are not met but the results are considered atypical (as observed from medical history and patient recall) then the patient can be re-screen on 1 occasion only.

Exclusion Criteria:

1. Women who are pregnant or breast feeding
2. Prior abdominal surgery which may cause bowel symptoms similar to IBS (note appendectomy and cholecystectomy will not be an exclusion)
3. Patients unable to stop anti-muscarinics, anti-spasmodics, high dose tricyclic antidepressants (i.e. above 50 mg/day), opiates/anti-diarrhoeal drugs*, NSAIDs (occasional over the counter use and topical formulations are allowed), long-term antibiotics, other anti-inflammatory drugs or 5-ASA containing drugs.
4. Patients on selective serotonin re-uptake inhibitors and low dose tricyclic antidepressants (i.e. up to 50 mg/day) for at least 3 months previous unwilling to remain on a stable dose for the duration of the trial.
5. Patients with other gastro-intestinal diseases including colitis and Crohn's disease.
6. Patients with the following conditions: Renal impairment, severe hepatic impairment or salicylate hypersensitivity.
7. Patients currently participating in another trial or have been in a trial within the previous 3 months
8. Patients who in the opinion of the investigator are considered unsuitable due to inability to comply with instructions
9. Patients with serious concomitant diseases e.g. cardiovascular, respiratory, neurological etc.

   * Loperamide is allowed as rescue medication through-out the trial, however if > 2 doses / week are taken during the screening phase then they are not eligible, though they can be re-screened on 1 occasion only.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average stool frequency during weeks 11 and 12. | Week 0 and week 12
  Clinical Endpoint
Change from baseline of number of mast cell per mm2 at week 12 | Week 0 and week 12
  Mechanistic endpoint

SECONDARY OUTCOMES:
Average daily severity of abdominal pain on a 0-10 scale | Week 0 to week 12
  Clinical Endpoint
Days with urgency | weeks 11-12
  Clinical Endpoint
Mean stool consistency using Bristol Stool Form Score | Week 0 to week 12
  Clinical Endpoint
Global satisfaction with control of IBS symptoms | Week 0 to week 12
  as assessed from the answer to the question "Have you had satisfactory relief of your IBS symptoms this week? Yes / No. "
Mast cell tryptase release during 6 hour biopsy incubation | Week 0 and week 12
  Mechanistic endpoint
IL-1β, TNF-a, histamine and serotonin secretion during same incubation | Week 0 and week 12
  Mechanistic endpoint
Small bowel tone assessed by volume of fasting small bowel water | Week 0 and week 12
  Mechanistic endpoint
Euro-Qol Score | Week 0 and week 12
  Ancillary endpoint
Centres for disease control and prevention health related quality of life healthy days core module score | Week 0 and week 12
  Ancillary endpoint
Hospital Anxiety Depression Scale Score | Week 0 and week 12
  Ancillary endpoint
Patient Health Questionnaire -15 | Week 0 and week 12
  Ancillary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Robin C Spiller, MD, Principal Investigator — NIHR Biomedical Research Unit, Nottingham University
Locations (1):
- Queen's Medical Centre, Nottingham, Notts, United Kingdom

REFERENCES:
- [Derived] Lam C, Tan W, Leighton M, Hastings M, Lingaya M, Falcone Y, Zhou X, Xu L, Whorwell P, Walls AF, Zaitoun A, Montgomery A, Spiller R. A mechanistic multicentre, parallel group, randomised placebo-controlled trial of mesalazine for the treatment of IBS with diarrhoea (IBS-D). Gut. 2016 Jan;65(1):91-9. doi: 10.1136/gutjnl-2015-309122. Epub 2015 Mar 12. PMID 25765462